CLINICAL TRIAL: NCT06835569
Title: A Phase 1/1b Multiple Cohort Trial of ALTA3263 in Patients With Advanced Solid Tumors With KRAS Mutations
Brief Title: A Study to Learn About Study Medicine ALTA3263 in Adults With Advanced Solid Tumors With KRAS Mutations
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alterome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3263-001
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Cancer; PDAC - Pancreatic Ductal Adenocarcinoma; NSCLC (Non-small Cell Lung Cancer); CRC (Colorectal Cancer); Advanced Solid Tumors
Keywords: KRAS mutation; NSCLC; Non-small cell lung cancer; Colorectal cancer; Pancreatic ductal adenocarcinoma; Colorectal carcinoma; Pancreatic cancer; Pancreatic carcinoma; Solid tumors; KRAS; Mutation; Metastatic; Advanced unresectable; Neoplasms; Neoplasms by Site; Carcinoma; Non-small cell lung carcinoma; Non-small cell lung neoplasm; Pancreatic neoplasm; Lung neoplasm; Colorectal neoplasm; Colon neoplasm; Mutant KRAS; KRAS amplification
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis; Neoplasms by Site; Carcinoma; Lung Neoplasms; Colonic Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ALTA3263 monotherapy (Experimental): ALTA3263 will be administered continuously at a protocol-defined dose based on cohort assignment
  Interventions: Drug: ALTA3263
- ALTA3263 in combination with cetuximab (Experimental): ALTA3263 in combination with cetuximab will be administered continuously at a protocol-defined dose based on cohort assignment
  Interventions: Drug: ALTA3263; Drug: cetuximab

INTERVENTIONS:
Drug: ALTA3263 — Oral ALTA3263 tablets will be administered at a protocol-defined dose
Drug: cetuximab — Cetuximab injection for IV use will be administered at a protocol-defined dose
  Arms: ALTA3263 in combination with cetuximab

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of ALTA3263 in adults with advanced solid tumors with KRAS mutations.

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 1/1b study of ALTA3263, an orally bioavailable KRAS isoform-selective inhibitor that inhibits multiple mutant forms of KRAS, in adults with advanced solid tumor malignancies with KRAS mutations. This study will evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary clinical activity of ALTA3263 as a monotherapy and as a combination regimen. The study consists of two parts: Part 1 - Dose Escalation and Part 1b - Dose Expansion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a solid tumor malignancy harboring a KRAS mutation identified through molecular testing (NGS- or PCR-based) with a Clinical Laboratory Improvement Amendments-certified (or equivalent) diagnostic test.
* Unresectable or metastatic disease.
* Progressed on, intolerant to, or declined prior standard-of-care therapy (including targeted therapy, if applicable) appropriate to tumor type and stage
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function

Exclusion Criteria:

* Prior treatment with a KRAS inhibitor, certain exceptions are described in the full study protocol
* Known condition that prohibits the ability to swallow or absorb an oral medication.

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Up to 39 months
  Number of participants that experience treatment-emergent adverse events (TEAEs).
Dose Limiting Toxicities | 21 days
  Number of participants with Dose Limiting Toxicities (DLTs).

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Cycle 1 (each cycle is 21 days) Day 1 (or Lead-in) and Day 15: Predose and up to 24 hours postdose
  Cmax
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Cycle 1 (each cycle is 21 days) Day 1 (or Lead-in) and Day 15: Predose and up to 24 hours postdose
  Tmax
Area Under Plasma Concentration Time Curve During the Dosing Interval (AUCt) | Cycle 1 (each cycle is 21 days) Day 1 (or Lead-in) and Day 15: Predose and up to 24 hours postdose
  AUCt
Terminal Half-Life (t1/2) | Cycle 1 (each cycle is 21 days) Lead-in phase: Predose and up to 48 hours postdose
  t1/2
Objective Response Rate (ORR) | Up to 39 months
  Assess per RECIST 1.1
Duration of Response (DOR) | Up to 39 months
  Assess per RECIST 1.1
Progression-Free Survival (PFS) | Up to 39 months
  Assess per RECIST 1.1
Overall Survival (OS) | Up to 39 months
  Assess per RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Study Medical Director, Study Director — Alterome Therapeutics
Locations (7):
- United States (7):
  - Research Site, Orlando, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No